CLINICAL TRIAL: NCT05603221
Title: Perfusion Assessment Using Arterial Spin Labelling MRI and Flat-panel Detector Parenchymal Blood Volume Imaging in Endovascular Treatment of Renal Artery Stenosis
Brief Title: Renal Perfusion Assessment in the Endovascular Treatment of Renal Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ASL and PBV in RAS
Record Dates: First submitted 2022-10-23; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Renal Artery Stenosis
Keywords: renal artery stenosis; renal perfusion
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endovascular Group: Patients who had successful endovascular revascularization

SUMMARY:
The clinical benefits of endovascular treatment in renal artery stenosis remain controversial. This study uses arterial spin labelling MRI and flat-panel detector parenchymal blood volume imaging to observe the change in renal perfusion after endovascular treatment in renal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who provided informed consent
* patients who were diagnosed with RAS by CTA, MRA, or Doppler ultrasonography
* patients who were aged 18 years or older
* patients whose intervened renal arteries were not completely occluded (confirmed by DSA)
* the stenosis percentage exceeding 70%
* patients who had uncontrolled blood pressure or impaired renal function
* paitents whose affected kidney did not have total loss of function

Exclusion Criteria:

* were pregnant
* had a history of renal transplantation or renal artery bypass surgery
* were allergic to iodine contrast medium
* had other contraindications of endovascular treatment
* contraindications of MRI examinations
* had technical failure in the endovascular treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted in renal artery stenosis patients aged 18 to 80 years with uncontrolled blood pressure or impaired renal function, who were intended for endovascular treatment. CTA, MRA, or Doppler ultrasonography were used for the assessment of the stenosis percentage of renal artery. Subjects with technical failure were excluded in order to reduce the influence of other variables.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Perfusion of the target kidney assessed by Arterial Spin Labelling MRI | Changes from baseline renal perfusion at 2 months
Perfusion of the target kidney assessed by Flat-panel Detector Parenchymal Blood Volume Imaging | Changes from baseline renal perfusion immediately after endovascular intervention

SECONDARY OUTCOMES:
Blood pressure | Changes from baseline blood pressure at 1 year
Renal function | Changes from baseline renal function at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China